CLINICAL TRIAL: NCT04924270
Title: Safety and Clinical Efficacy Associated With Faecal Microbiota Transplantation Performed in Treatment-naïve Patients With Newly Diagnosed Rheumatoid Arthritis, Ankylosing Spondylitis, Psoriatic Arthritis, Pulmonary Sarcoidosis, Crohn's Disease, and Ulcerative Colitis: a 52-week, Double-blind, Randomised, Placebo-controlled, Exploratory Trial
Brief Title: Safety and Efficacy of Capsule FMT in Treatment-naïve Patients With Newly Diagnosed Chronic Inflammatory Diseases
Acronym: FRONT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Region of Southern Denmark (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Torkell Ellingsen, MD PhD, Clinical professor and head of research, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20/3106
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis; Ankylosing Spondylitis; Psoriatic Arthritis; Crohn Disease; Ulcerative Colitis
Keywords: Faecal microbiota transplantation; Fecal microbiota transplantation
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic; Crohn Disease; Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cFMT (Experimental)
  Interventions: Biological: Faecal microbiota transplantation
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Faecal microbiota transplantation — The capsule FMT transplant consists of faeces obtained from a thoroughly screened, unpaid, anonymous stool donor. Each FMT product is made from 50g faeces diluted in sterile saline (0.9% NaCl) and glycerol, blended, centrifuged and filtered to remove particulate material before transfer to double-layered capsules. The FMT capsules will be stored at - 80 ⁰C until use. On the day of the FMT, the FMT capsules will be thawed to room temperature before treatment.
  Other Names: capsule FMT
  Arms: cFMT
Other: Placebo — Placebo capsules consist of NaCl (0.9%) and glycerol added brown food colouring.
  Arms: Placebo

SUMMARY:
PURPOSE: The main purpose is to explore clinical efficacy and safety associated with capsule FMT (cFMT) performed in newly diagnosed, untreated patients with rheumatic and gastrointestinal chronic inflammatory diseases (CIDs).

DESIGN AND METHODS: In this 1:1 double-blind, placebo-controlled, randomised, 12-month exploratory trial, 200 patients with at least one of 6 different diagnoses of CIDs fulfilling the study criteria will be enrolled at time of diagnosis. The patient groups are: rheumatoid arthritis (RA), ankylosing spondylitis (AS), psoriatic arthritis (PsA), Crohn's disease (CD), and ulcerative colitis (UC). The primary endpoint is change from baseline to eight weeks in the physical component summary (PCS) of the short form health survey (SF-36). Key secondary clinical endpoints will be evaluated at 8 weeks. Other secondary clinical endpoints will be evaluated at 52 weeks and reported in secondary papers.

The baseline visit will be performed as quickly as possible after the patient's informed consent has been obtained to ensure no unnecessary treatment delay. Stratified by CID diagnosis, patients will be randomised (1:1) to either placebo or single-donor cFMT processed from stool provided to the hospital from anonymous-to-the-patient healthy donors. The experimental intervention FMT/placebo will be repeated once weekly the first month (i.e., each patient will receive a total of four treatments). In addition, all participants will concomitantly be offered the national guideline first-line anti-inflammatory treatment following the baseline visit.

At baseline, 8 weeks, 26 weeks, and 52 weeks a thorough clinical examination will be conducted and all relevant clinical scores for each disease entity will be registered. Patient-reported-outcomes including SF-36 and disease specific questionnaires will be collected at week 1, 2, 3, 4, 8 (primary endpoint evaluation), 26 and 52. Adverse events will be monitored through out the trial.

ELIGIBILITY:
Inclusion criteria:

* Newly diagnosis of treatment-naïve RA, AS, PsA, PSar, CD, or UC.
* Treatment-naïve which is defined as no current or previous (within 3 months) disease-modifying anti-rheumatic drugs (DMARDs) or systemic anti-inflammatory treatment including glucocorticoids.
* Presence of CID treatment indication (no contra-indications) and patient accept to start first-line standard treatment in accordance with the national guideline for the specific diagnosis following the baseline visit.
* Age 18 to 75 years.

Exclusion criteria:

* Indication for biological therapy as primary therapy.
* Celiac disease or food allergy.
* Current cancer.
* Hepatitis B and C, HIV, HTLV1/2, and active TB or other serious chronic infections.
* Pregnant or breastfeeding women.
* Not wishing to participate or not suited for FMT intervention or project evaluation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical Component Summary score (PCS) | 8 weeks (+/- 1 week)
  Change from baseline in the Physical Component Summary score (PCS) of the 36-Item Short Form Health Survey (SF-36)

SECONDARY OUTCOMES:
Treatment failure | 8 weeks (+/- 1 week)
  Proportion of patients experiencing treatment failure at 8 weeks
Mental Component Summary score (MCS) | 8 weeks (+/- 1 week)
  Change from baseline in the Mental Component Summary score (MCS) of the 36-Item Short Form Health Survey (SF-36)
Physician's Global Assessment | 8 weeks (+/- 1 week)
  Change from baseline in the Physician's Global Assessment (0-100 mm VAS)
Patient's Global Assessment | 8 weeks (+/- 1 week)
  Change from baseline in the Patient's Global Assessment (0-100 mm VAS)
Fatigue | 8 weeks (+/- 1 week)
  Change from baseline in Fatigue visual analogue scales (0-100 mm VAS)
C-reactive protein | 8 weeks (+/- 1 week)
  Change from baseline in C-reactive protein

OTHER OUTCOMES:
Other secondary endpoints, specific for each disease | 8 weeks (+/- 1 week)
  Disease specific outcomes, not mentioned above
Tertiary (secondary exploratory) endpoints | 52 weeks (+/- 2 weeks)
  All of the above efficacy outcomes and safety outcomes assessed after 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Torkell Ellingsen, MD PhD, Principal Investigator — Odense University Hospital; Maja S Kragsnaes, MD PhD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request. This will require review and approval by the trial scientific board and the data responsible parties. Terms of collaboration will be reached together with a signed collaboration agreement and data processor agreement.
Supporting Information: Study Protocol, SAP